CLINICAL TRIAL: NCT04641806
Title: Clinical and Immunological Evolution of Covid-19 Occurring in a Context of Non-Hodgkin Lymphoma
Acronym: LYMPHO-Cov-2
Status: Withdrawn | Type: Observational
Why Stopped: Following submission of the amended protocol, the ethic commitee requested sponsor to resubmit it like a new protocol
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Caroline BESSON, Investigator Coordinator, Versailles Hospital
Other Study IDs: P20/21_LYMPHO-Cov-2
Record Dates: First submitted 2020-11-20; First posted 2020-11-24 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: B-cell Lymphoma; Covid19
MeSH Terms: conditions — Lymphoma, B-Cell; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples from cases and controls
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lymphoma cases: Adults aged at least 18 years, with a Covid-19 confirmed by PCR, diagnosed between February and May 2020. Past history of B-cell NHL in remission, active surveillance or during first-line or second-line treatment Affiliated with a social security, consenting to the study
- Controls: Adults aged at least 18 years, with a Covid-19 confirmed by PCR, diagnosed between February and May 2020. No past history of lymphoma .
  Affiliated with a social security, consenting to the study

SUMMARY:
France was gradually affected by SARS-Cov-2 from January 2020; it evolved in an epidemic mode in March and April 20. During the 1st phase of the epidemic, more than 250 000 cases of Covid-19 have been confirmed in France resulting in the death of more than 30,000 patients. Mortality from infection varies greatly depending on the age of the affected individuals and their comorbidities including a history of cancer. We conducted a retrospective study in 89 patients with lymphoma and Covid-19 during the first phase of the epidemic and showed a 30-day mortality of 29%. Mortality was higher in patients over 70 years of age and in a situation of relapsed or refractory disease. Lymphoma-induced hypogammaglobulinemia and / or lymphopenia as well as chemotherapy and immunotherapy treatments are known to promote the development of infections in affected individuals. Among these, anti-CD20 monoclonal antibodies, widely prescribed to treat B-cell non-Hodgkin lymphomas (B-NHL) induce a rapid depletion of over 95% of mature CD20 + B cells. This can alter the production of antibodies, and the constitution of memory responses to a new pathogen. Also, B lymphocytes have a key immunomodulatory role in the control of viral infections.

The specific immune response to SARS-CoV -2 and its evolution remain under characterization. Regardless of their neutralizing capacity, specific IgM appear 5 days after the onset of symptoms while IgG appear after 14 days. The immune response to SARS-CoV-2 also includes a T lymphocyte component, with an increase, among circulating lymphocytes, of activated CD8 and CD4 T lymphocytes. Data are still lacking on the specific response of CD4 and CD8 T lymphocytes against SARS-CoV-2, but these responses probably play a crucial role in virus clearance as well as in the immunopathology associated with SARS-CoV-2. Therapeutic depletion of B lymphocytes before acute infection may alter the generation of primary and functional responses. Therefore, a growing concern is whether patients with B-NHL who have acquired an infection with SARS-CoV-2 are protected against re-infection in the same way when they have or have not received anti-CD20 monoclonal antibodies.

Analyzing the clinical and immunological evolution of Covid-19 in patients with B-NHL is useful to adapt the treatment recommendations in their regard according to the risk of severe form of Covid-19 . This is a multicenter, prospective study to determine whether treatment with monoclonal anti-CD20 antibodies in patients with B-cell NHL modifies the clinical and immunological course of Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* adults aged at least 18 years
* Covid-19 confirmed by PCR
* between February and May 2020
* affiliated with a social security
* consenting to the study

Case specific inclusion criteria :

* being or having been affected by B-NHL
* being currently in remission, active surveillance or during first-line or second-line treatment

Exclusion Criteria:

* Subjects less than 18 years old
* Subject with protective measure (curatorship, guardianship, safeguard of justice) -Subjects unable to give consent
* Pregnant or breastfeeding women
* Subject refusing to participate
* Case-specific non-inclusion criteria :
* Patient with a life expectancy linked to NHLof less than 6 months or with a History of hematopoietic allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient recruitment will be done from the hematology units of the 10 centers. The recruitment of controls will be done from the spouses of the patients. A number of 100 case patients and 20 controls is to be recruited during the 4-month inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Immunological response to SARS Cov2 | 6 months to one year ater Covid-19
  Quantification of IgG anti-SARS-Cov-2 by ELISA.
Clinical evolution after Covid-19 diagnosis | 6 months after Covid-19
  length(s) of stay(s) for Covid-19 in hospitalization and intensive care

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lamure S, Dulery R, Di Blasi R, Chauchet A, Laureana C, Deau-Fischer B, Drenou B, Soussain C, Rossi C, Noel N, Choquet S, Bologna S, Joly B, Kohn M, Malak S, Fouquet G, Daguindau E, Bernard S, Thieblemont C, Cartron G, Lacombe K, Besson C. Determinants of outcome in Covid-19 hospitalized patients with lymphoma: A retrospective multicentric cohort study. EClinicalMedicine. 2020 Oct;27:100549. doi: 10.1016/j.eclinm.2020.100549. Epub 2020 Oct 13. PMID 33073216